CLINICAL TRIAL: NCT07107165
Title: Adapting After Discharge From Allogeneic SCT: Partnering Together; Dyadic Intervention to Improve Patient-Family Caregiver Team-Based Management of the Medical Regimen After Allogeneic Hematopoietic Cell Transplantation
Brief Title: Psychosocial and Behavioral Intervention for Stem Cell Transplant Patients and Their Family Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Donna Posluszny, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: STUDY25020163; R01CA268004 (NIH)
Record Dates: First submitted 2025-07-17; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Stem Cell Transplant; Hematopoetic Stem Cell Transplant; Hematopoetic Stem Cell Transplantation
Keywords: stem cell transplant; hematopoietic stem cell transplant
MeSH Terms: interventions — 1-(di-(2-pyridyl)methylene)-5-salicylidenethiocarbonohydrazide; Palliative Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dyadic Problem Solving Training (DPST) (Experimental): DPST will teach problem solving skills to both the patient and family caregiver as they manage the medical regimen.
  Interventions: Behavioral: Dyadic Problem Solving Training
- Supportive Care (Active Comparator): Supportive Care will provide support to both the patient and family caregiver as they manage the medical regimen.
  Interventions: Behavioral: Supportive Care

INTERVENTIONS:
Behavioral: Dyadic Problem Solving Training — DPST consists of teaching the patient and family caregiver problem-solving skills that they can apply to help them manage the medical regimen after stem cell transplant.
  Other Names: DPST
  Arms: Dyadic Problem Solving Training (DPST)
Behavioral: Supportive Care — Supportive Care consists of providing support to the patient and family caregiver as they manage the medical regimen after stem cell transplant
  Other Names: SC
  Arms: Supportive Care

SUMMARY:
Adherence to the medical regimen after stem cell transplant is challenging for both patients and their family caregivers. The investigators propose a randomized clinical trial testing two brief psychosocial interventions to determine if either improves patient and family caregiver psychosocial and health-related outcomes.

DETAILED DESCRIPTION:
The investigators propose a randomized controlled trial testing two brief, 4 session psychosocial interventions to help patients and family caregivers better manage the time period after hospital discharge from stem cell transplant. Patients and family caregivers will be randomized to either the skill learning intervention (n=52 patient-family caregiver dyads) or to the supportive care intervention (n=52 patient-family caregiver dyads). The intervention will be conducted via live video conferencing. Patients and family caregivers will complete questionnaires before the intervention and at 1-, 5-, 12-, 24 weeks afterwards. The investigators will determine whether the skills learning group has improved outcomes, including adherence to the medical regimen and perceived task efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for stem cell transplant at the University of Pittsburgh Hillman Cancer Center
* 18 years or older
* having a family caregiver age 18 years or older also willing to participate in the study
* willing to accept randomization

Exclusion Criteria:

* Prior history of stem cell transplant
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Health Habits Assessment - modified for stem cell transplant | 1-, 5-, 12- and 24-weeks post-intervention
  Assess levels of adherence to the post-transplant multi-component medical regimen of 20 main tasks; each task marked as yes = 1/no=0 adherent. Tasks will be grouped and summed into categories including medication taking (3 items, range 0=low to 3 high), infection precautions (6 items; range 0=low to 6 high), catheter/port care (4 items, range 0=low to 4 = high), and lifestyle behaviors (7 items, range 0=low to 7=high). Higher scores indicate greater adherence.
Perceived task efficacy | 1-, 5-, 12- and 24-weeks post intervention
  Assesses perceptions of efficacy to complete tasks of the post-transplant multi-component medical regimen, 20 items rated on 1=low to 10=high scale, mean score will be used.

SECONDARY OUTCOMES:
Immunosuppressant blood levels | 1-, 5-, 12- and 24-weeks post-intervention
  levels of immunosuppressant medication in patient's blood
Patient health care utilization | continuous over 24 weeks post-intervention
  Counts of number of hospital readmissions, emergency room visits, and unplanned medical visits
Patient Health Questionnaire- 9 | baseline and 1-,5-,12-, and 24-weeks post-intervention
  Assesses symptoms of depression, 9 items rated on 4-point scale from 0=not at all to 3=nearly every day. Sum and categorical classification will be used (score 10-14=moderate; score 15 and higher =severe.
Generalized Anxiety Disorder - 7 | baseline and 1-, 5-, 12-, and 24-weeks post-intervention
  Assesses symptoms of anxiety, 7 items rated from 0=not at all to 3=nearly every day. Sum and category will be used (score 10-14 = moderate; score 15 or higher = severe)
Dyadic Adjustment Scale - modified | baseline and 1-, 5-, 12-, 24-weeks post-intervention
  Assess relationship quality, 9 items rated from 1=not at all to 5 = often; range 9-45; sum will be used. Higher scores indicate greater relationship quality.
Task Responsibility | 1-, 5-, 12-, and 24-weeks post-intervention
  Rating of whether the patient was mostly responsible, the caregiver was mostly responsible, or the patient and caregiver had equal responsibility in making sure each task of the post-transplant multi-component medical regimen is completed. Levels of each of the three choices will be tabulated. The highest level will dictate the categorical score (patient mostly responsible; caregiver mostly responsible; patient and caregiver equally responsible).
Caregiver Reaction Assessment | 1-, 5-, 12-, 24- weeks
  Assesses burden in caregivers, 24 items rated on a 1=low to 5=high; range = 24-120; sum will be used.
Cancer and Treatment Distress Scale | baseline and 1-, 5-, 12-, 24-weeks post-intervention
  Assess distress specific to cancer, 35 items are rated from 0=none to 3=severe; range = 0-105; sum score will be used.
PROMIS - 16 v2.1 | baseline and 1-, 5-, 12-, and 24-weeks post-intervention
  Assesses overall health-related quality of life and functioning, 16 items rated from 1=low to 5 = high; higher scores indicate greater health-related quality of life; sum will be used.

OTHER OUTCOMES:
Client Satisfaction Assessment - 8 | 1-week post intervention
  Ratings of satisfaction with the intervention, 8 items, rating scale from 1 (low) to 4 (high). Sum of ratings on each item will be used with higher scores indicating greater satisfaction.
Satisfaction with Telehealth Technology | 1-week post intervention
  assess satisfaction with telehealth services, 2 items rated on 1=low to 7=high scale range = 2-14; sum will be used.
clinical outcomes | continuous over 24-weeks post-intervention
  presence of graft failure, graft versus host disease, and survival
Lack of Attention from Health Care Professionals | 1-, 5-, 12- and 24-weeks post-intervention
  A four-item subscale of the Cancer Caregiving Tasks, Consequences of Needs scale. Items have five possible responses: always/most days = 4; mostly=3; only sometimes=2; rarely/never=1, and don't know/not relevant=0. Items are summed to make a total score; higher score indicates more attention from health care professionals.
Worry about mistakes | 1-, 5-, 12- and 24-weeks post-intervention
  1 item specifying how worried are you about making a mistake or unintentionally hurting the patient while caring for him/her. Responses include 1=very worried; 2=somewhat worried; 3=only a little; 4=not at all. Lower responses indicate greater worry.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh Medical Center Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The study database will be reviewed to ensure that no identifying information of any type is contained therein. A downloadable, de-identified data set and data dictionary will be made available electronically from the PI after the request is reviewed by the research team for scientific merit and requestors provide evidence to the PI that (a) their plan for the use of such data has been approved by their institution's Institutional Review Board or its equivalent, and (b) they have completed NIH requirements for training in research integrity and human subjects protection.
Supporting Information: Study Protocol, SAP
Time Frame: To provide the investigators adequate time to prepare and submit the majority of publications likely to result from the research, data obtained from the study will be made publicly available no sooner than 18 months after the conclusion of the study.
Access Criteria: Access can be requested from PI following plan description and time frame noted above

REFERENCES:
- [Background] Posluszny DM, Bovbjerg DH, Syrjala KL, Agha M, Dew MA. Correlates of anxiety and depression symptoms among patients and their family caregivers prior to allogeneic hematopoietic cell transplant for hematological malignancies. Support Care Cancer. 2019 Feb;27(2):591-600. doi: 10.1007/s00520-018-4346-3. Epub 2018 Jul 19. PMID 30022348
- [Background] Posluszny DM, Bovbjerg DH, Syrjala KL, Agha M, Farah R, Hou JZ, Raptis A, Im AP, Dorritie KA, Boyiadzis MM, Dew MA. Rates and Predictors of Nonadherence to the Post-Allogeneic Hematopoietic Cell Transplantation Medical Regimen in Patients and Caregivers. Transplant Cell Ther. 2022 Mar;28(3):165.e1-165.e9. doi: 10.1016/j.jtct.2021.11.020. Epub 2021 Dec 4. PMID 34875403